CLINICAL TRIAL: NCT01011985
Title: A Study of the Effect of Hemodialysis Access Type on Markers of Inflammation
Brief Title: A Study Evaluating the Association of Inflammation With Hemodialysis Access Type
Status: Completed | Type: Observational
Sponsor: Montefiore Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: 06-07-336E
Record Dates: First submitted 2009-11-09; First posted 2009-11-11 (Estimated); Last update posted 2018-07-09 (Actual); Status verified 2018-07

CONDITIONS: End Stage Renal Disease; Inflammation
Keywords: end stage renal disease; inflammation; vascular access; hemodialysis
MeSH Terms: conditions — Kidney Failure, Chronic; Inflammation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — serum
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- AVF: Initial access is an AVF
- AVG: Initial vascular access is an AVG
- TC: Initial vascular access is a tunneled catheter, with or without a maturing AVF or AVG

SUMMARY:
To determine if the type of hemodialysis vascular access correlates with markers of inflammation, namely C-reactive protein and interleukin-6, and with both access and patient survival in the end stage renal disease population.

DETAILED DESCRIPTION:
A Study Of The Effect Of Hemodialysis Vascular Access Type On Markers Of Inflammation PI: Michele H. Mokrzycki MD, MS

Introduction/Background: The prevalence of chronic inflammation is high (35-65%) in end stage renal disease (ESRD) patients and is associated with an increased risk of atherosclerosis, and overall and cardiovascular mortality in this population.(1-4) Stenvinkel et al observed that a pre-HD C-reactive protein (CRP) level of >10 was associated with a higher prevalence of carotid plaques (p<0.01), and clinical manifestations atherosclerotic cardiovascular disease (MI, CVA, PVD) (p<0.05) in the ESRD population. (1) Zimmerman et al report a 2.7-fold and 4.6-fold higher risk of 2 yr all-cause mortality associated with a CRP level between 7.5-15.7. and >15.7, respectively. The cardiovascular mortality was similar (2.9-fold, and 5.5-fold). A single elevated CRP level has been shown to be a powerful indicator of mortality in ESRD patients, even after 4-5 years of follow-up. (3).

CRP is a sensitive major acute phase protein, synthesized by hepatocytes under transcriptional control by IL-6. In the presence of human serum, CRP induces the expression of MCP-1, VCAM-1, ICAM-1, and E-selectin. (5). The interaction of CRP with monocytes in vitro results in the release of IL-1 β, IL-6, TNF-α, and tissue factor.(6)

The origin of inflammation in the ESRD population is unclear, although the HD session per se has been implicated. Korevaar et al studied the effect of the HD session on CRP level and mortality in 186 pts. (7) Thirty-eight % of patients had a CRP level below detection (<3 mg/L), and in those patients with detectable CRP levels pre-HD 37% had no increase with HD, and 25% of patients had an increase (mean +2.3 (0.6-9.2)) in CRP level (adjusted for change in blood volume) during HD. There was no difference in pre-HD CRP level between the latter 2 groups. A lower 2 yr survival was observed in the group in which CRP increased during HD, (44 vs. 66%, p=0.09). After adjusting for nutritional factors, age, comorbidity and primary kidney disease, a rise of 1 mg/dl in CRP during a HD session, was associated with an increase in mortality risk of 9% (Adjusted hazard ratio 1.09, 95%CI=1.09-1.16) Independent predictors of high CRP levels during HD include patient age (β=0.07, p=0.05), pre-HD CRP (β=0.95, p<0.01), 2 needle dialysis (β=2.39, p=0.05, and cholesterol ((β= -0.92, p=0.04).

Additional possible reasons for increased markers of inflammation in the ESRD population include 1) uremia-related alterations in immune/host defense systems, specifically increased cytokine production, 2) increased oxidative stress (oxidized-LDL), advanced glycation end products (AGEs) 3) the dialysis membrane (IL-6 and IL-1 β production by certain membranes), 4) contaminated dialysate, [ultrapure dialysate reduces CRP levels],5) intercurrent clinical events, 6) and occult arteriovenous graft infection, 7) protein-energy malnutrition, and 8) shorter time on hemodialysis (HD). (8-13). None of the above CRP associated mortality studies controlled for type of vascular access. There are reports of an association of vascular access type with other markers of inflammation. Kaysen et al report an association between low levels of serum albumin with presence of an AVG, and Thadani et al recently reported elevated WBC count and hemocatheters (14,15).

Polkinghorne et al studied the effect of vascular access in incident hemodialysis patients on all-cause mortality using multivariate analysis.(16) In this adjusted analysis, catheter use and AVGs were associated with significant excess mortality. Compared to AVFs, catheters were associated with a 3.3-fold higher and AVGs with a 1.6-fold higher all-cause mortality after 120 days. However, the authors speculate that, in part, this may due to the higher risk of infections. In fact the risk of infectious death was 1.7-fold higher with AVGs, and 2.7 fold higher with catheters. The risk of the type of vascular access with inflammation, independent of infection, is unknown.

Research Question/Objective: To determine if the type of HD vascular access correlates with markers of inflammation, namely CRP and IL-6, and with both access and patient survival in the ESRD population.

Study Design: A prospective study using a multiple group design.

Subjects: Incident ESRD patients. Patients with Stage IV and V (GFR <30 ml/min using MDRD mod equation) will be recruited from the renal clinics and private practices. Sites include both the Moses and Weiler campuses of the Montefiore Medical Center in Bronx, NY. Type of vascular access to be inserted will be determined on clinical grounds by the patient's nephrologist and access surgeon, these include hemocatheter, arteriovenous graft, and arteriovenous fistula.

Study Procedures: Blood samples (10 cc) will be drawn immediately (within 24 hours) prior to access surgery, and 1 week, and 1, 3, 6 and 12 months, and upon dialysis initiation.(6 samples per subject over 1 year) Once the patient is on hemodialysis the blood samples will be drawn pre-HD via the access. Samples will be centrifuged immediately (3000 rpm x 10 minutes), cooled within 1 hour, and stored at -80 degrees C. Pre-dialysis samples will be tested for high-sensitivity C-Reactive Protein (hsCRP) TNF-α and IL-6 (both ELISA assay, plasma by sandwich-type immunoassay) levels. Patient demographic and other clinical data will be recorded, This includes age, race, sex, body surface area, DM, SLE and other connective tissue diseases, malignancy, history of atherosclerotic diseases (CAD, PVD, CVA), active infection, history of viral infection with hepatitis B or C, human immunodeficiency virus. Routine monthly lab results drawn pre-dialysis as part of clinical practice will be recorded, these include serum albumin, complete blood count, electrolytes, blood urea nitrogen, creatinine, liver function tests, and lipid profile. Medications will be reviewed for the presence of ACE-Inhibitors, ARBs, aspirin, NSAIDS, statins. A subjective global assessment score (SGA) and comorbidity risk score will be performed. (17,18) Date of HD initiation, and type of HD membrane will be recorded. Clinical events after vascular access surgery will be monitored, including infection, hospitalization (reason), MI, CVA. Outcomes to be recorded will include access survival (primary and secondary patency), patient mortality (all-cause, infectious and cardiovascular).

Data Management and Analysis: Differences in hs-CRP, TNF-α and IL-6 levels between the 3 vascular access groups for all time periods (baseline, 1 week, 1, 3, 6,12 months) will be analyzed using a random effects (mixed) model, with time as a random effect. A Power analysis was performed by Kathrine Freeman, PhD in the Department of Biostatistics and Epidemiology at Montefiore Medical Center, using multiple comparisons between groups. We hypothesize a 100% increase in hsCRP level from baseline in the catheter group and a 10% increase in the AVF group. We predict that the AVG group will have an increase in hs CRP between 10-100%. The initial power analysis (80%, 2-tailed α=0.05) predicted that 51 subjects per group would be needed. Anticipating a 20% dropout rate per year, we will recruit 61 subjects will be required in each group. All hsCRP data will be transformed, most likely using a log scale, as per prior studies and upon review of the distribution of the data. Dunnett's multiple comparison procedure will be performed for the 2 contrasts (each group, ie. the AVF and AVG groups, compared with the tunneled catheter group. A multivariate analysis using a mixed effects model will be performed to determine the factors related to a change in CRP level at baseline and at 1 week, 3, 6, 12 months. Patient and access survival will be analyzed using Kaplan-Meier method and Cox proportional hazards regression analysis.

Blood specimens will be stored in a -70 freezer in Dr. Joel Neugarten's lab, Moses 6th floor laboratories. Patient charts will be coded and stored in a locked file cabinet in Dr. Mokrzycki's office, Centennial 4th floor at Montefiore Medical Center. One of the co-investigators will perform the sandwich immunoassays for hsCRP, TNF-α and IL-6 in Dr. Victor Schuster's lab, Ullman Building 6th floor.

Implementation plan/timetable: Enrollment of subjects by Dr. Mala Sachdeva, and Peter Durkin, PA will begin once the protocol has been approved by the IRB. The sites of patient identification and enrollment, and baseline specimens will be the Renal Clinics at Montefiore and Weiler Hospitals, and from the Renal Faculty practices. Follow-up specimens will be drawn at the above sites, while the patients are pre-hemodialysis, and will be drawn before the dialysis session for patients already receiving hemodialysis. Both preliminary and follow-up data entry will be performed by Dr. Mala Sachdeva using SPSS. Patient charts/records and specimens will be coded to ensure confidentiality. Specimens and charts will be stored as described above. Data analysis will be performed by Dr. Mokrzycki, Dr. Sachdeva and Dr Kathrine Freeman. The anticipated duration of the study is 3 years: approximately 2 years for patient enrollment and 1 year of follow-up data and time for data analysis.

ELIGIBILITY:
Inclusion Criteria:

* CKD patients referred for their initial vascular access
* Able to consent for surgery/study

Exclusion Criteria:

* Active inflammatory states
* Active infection
* Autoimmune diseases
* Acute renal allograft rejection
* HIV positive status

Ages: 18 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Incident stage 4 and 5 chronic kidney disease patients receiving their first dialysis access.
Sampling Method: Probability Sample
Enrollment: 64 (Actual)
Dates: Start 2006-08; Primary Completion 2008-04 (Actual); Study Completion 2008-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michele H Mokrzycki, MD, MS, Principal Investigator — Montefiore Medical Center
Locations (1):
- Montefiore Medical Center and Jack D Weiler Hospital, The Bronx, New York, United States